CLINICAL TRIAL: NCT06474156
Title: Motiv8: Examining Treatment Motivation Among Youth and Parents in Forensic Treatment
Brief Title: MOTIV8 - Treatment Motivation in Forensic Youth Treatment
Status: Recruiting | Type: Observational
Sponsor: University of Amsterdam (Other)
Collaborators: Kwaliteit Forensische Zorg Jeugd (Unknown)
Responsible Party: Principal Investigator, Jet Westerveld, MSc., University of Amsterdam
Other Study IDs: JWesterveld
Record Dates: First submitted 2024-06-05; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Motivation
Keywords: Treatment Motivation; Multidimensional Family Therapy; Youth; Parents; Delinquency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- short-stay residents juvenile justice center: For the first group (first series case studies), ten short-stay residents will be included who enter residential MDFT and, after 1-3 months in the facility, continue MDFT on an outpatient basis.
  MDFT is a systemic intervention for juveniles and young adults exhibiting delinquent behavior and/or experiencing disorders related to alcohol and/or drug use. MDFT for short-term residents is indicated by a behavioral scientist following multidisciplinary consultation if there are serious concerns about the parent-child relationship and/or the family situation
  Interventions: Behavioral: Multidimensional Family Therapy
- long-stay residents juvenile justice center: For the second group (second series of case studies), six long-term residents will be included. For long-term residents, MDFT is routinely recommended, provided that the inclusion criteria are met.
  Interventions: Behavioral: Multidimensional Family Therapy

INTERVENTIONS:
Behavioral: Multidimensional Family Therapy — Multidimensional family therapy is a manualized,evidence-based, intensive intervention program with assessment and treatment modules focusing on four areas: (a) the individual adolescents' issues regarding substance use disorder, delinquency, and comorbid psychopathology, (b) the parents' child-rearing skills and personal functioning, (c) communication and relationship between adolescent and parent(s), and (d) interactions between family members and key social systems (Liddle, 2002).
  Other Names: MDFT

SUMMARY:
This project entails to gain a deeper understanding of the development of treatment motivation over the course of intramural and outpatient forensic youth care. Research questions are 1) How does treatment motivation of youth and parents develop over the course of forensic systemic therapy, and following the transition from inpatient to outpatient therapy?; 2) Which client factors, interpersonal factors, and contextual characteristics moderate the development of treatment motivation?; 3) Which mechanisms play a role in the development of treatment motivation?; and 4) How does treatment motivation affect treatment retention and the achievement of primary therapy goals?

DETAILED DESCRIPTION:
Multidimensional Family Therapy (MDFT) has been shown to motivate youth and parents in forensic care for treatment. The current study will investigate the development of treatment motivation of youth and parents over the course of MDFT, offered in a juvenile justice center. Furthermore, mechanisms and moderators will be examined, in addition to the impact of treatment motivation on treatment retention and goal achievement. Two studies with a Multiple Case Experimental Design (MCED), one with an ABC design (A = baseline, B = residential MDFT, and C = outpatient MDFT) and one with an AB design, will be conducted. Juveniles who enter residential MDFT, during a short detention period (study 1; 10 cases) or during a longer detention period (study 2; 6 cases) will be recruited, as will their parents.

ELIGIBILITY:
Inclusion Criteria:

- entering residential MDFT

Exclusion Criteria:

- (only for short term residents) residing more than an hours' drive from the juvenile justice center after detention

Ages: 12 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Residents in a juvenile justice center
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Treatment motivation youth perspective (validated questionnaires) | at least 5 times during phase A (2-6 weeks); every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Treatment Motivation Questionnaire for Adolescents (van der Helm et al., 2013; van der Helm et al., 2018; 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree), with a higher score indicating more motivation for treatment; Cooperation Scale (Tolan et al., 2002; 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree. A higher total score indicates more motivation for treatment).
Treatment motivation caregiver perspective (validated questionnaires) | at least 5 times during phase A (2-6 weeks); every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Parent Motivation Inventory (Nock & Photos, 2006); Cooperation Scale (Tolan et al., 2002). Participants respond on a 5-point Likert scale on both questionnaires ranging from 1 (completely disagree) to 5 (completely agree). Higher total scores indicate more motivation for treatment.
Treatment motivation therapist perspective (validated questionnaires) | every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Cooperation Scale (Tolan et al., 2002; 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates more motivation for treatment).
Treatment motivation (qualitative data) | Youth/Caregivers: at the end of each phase (A (after 2-6 weeks), B (after 1-9 months) and C (after 1-3 months))
  Youth/Caregivers: semi-structured interview

SECONDARY OUTCOMES:
Therapeutic alliance youth perspective | every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Session Rating Scale (SRS; Duncan et al., 2003). The SRS is scored by adding the total of the client's marks on the four 10-cm lines, with a higher total score indicating a stronger alliance.
Therapeutic alliance caregiver perspective | every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Session Rating Scale (Duncan et al., 2003). The SRS is scored by adding the total of the client's marks on the four 10-cm lines, with a higher total score indicating a stronger alliance.
Sense of competence youth perspective | at least 5 times during phase A (2-6 weeks); every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Basic Psychological Need Satisfaction and Frustration Scale (Chen et al., 2015), subscales Competence Satisfaction and Competence Frustration. Participants respond on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). A higher total score indicates a higher sense of competence.
Sense of competence caregiver perspective | at least 5 times during phase A (2-6 weeks); every other week during phase B (1-9 months; at least 5 assessments), at least 5 times during phase C (1-3 months).
  Basic Psychological Need Satisfaction and Frustration Scale (Chen et al., 2015), subscales Competence Satisfaction and Competence Frustration. Participants respond on a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). A higher total score indicates a higher sense of competence.
Aggression and rule-breaking behavior youth perspective | The complete subscale is administered in phase A (2-6 weeks), every other week during phase B (1-9 months) and C (1-3 months) the (3-5) items reflecting the most severe problems are selected.
  Youth Self Report (YSR; Achenbach, 1991), subscale aggression and rule-breaking behavior. Youth complete the YSR by rating their behavior on a three-point scale for the 30 items in this subscale. Specifically, the child rates the behavioral symptoms as '0' if not present, a '1' if the child sometimes exhibits the symptom and '2' if the child frequently demonstrates the symptom. A higher total score indicates more aggression and rule breaking behavior.
Aggression and rule-breaking behavior caregiver perspective | The complete subscale is administered in phase A (2-6 weeks), every other week during phase B (1-9 months) and C (1-3 months) the (3-5) items reflecting the most severe problems are selected.
  Child Behavior Checklist (CBCL; Achenbach, 1991), subscale aggression and rule-breaking behavior. Parents complete the CBCL by rating their children on a three-point scale for the 30 items in this subscale. Specifically, a parent rates the behavior as a '0' if it is not present, a '1' if the child sometimes exhibits the symptom, and a '2' if the child frequently demonstrates the symptom. A higher total score indicates more aggression and rule breaking behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- JJC Teylingereind, Sassenheim, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the sensitive nature of the data, they will not be made publicly available.

REFERENCES:
- [Background] Duncan, B. L., Miller, S. D., Sparks, J. A., Claud, D. A., Reynolds, L. R., Brown, J., & Johnson, L. D. (2003). The Session Rating Scale: Preliminary psychometric properties of a "working" alliance measure. Journal of brief Therapy, 3(1), 3-12.
- [Background] Chen, B., Vansteenkiste, M., Beyers, W., Boone, L., Deci, E. L., Van der Kaap-Deeder, J., ... & Verstuyf, J. (2015). Basic psychological need satisfaction, need frustration, and need strength across four cultures. Motivation and Emotion, 39, 216-236. https://doi.org/10.1007/s11031-014-9450-1
- [Background] Achenbach, T. M. (1991b). Manual for the Youth Self-Report and 1991 Profile. Burlington: University of Vermont, Department of Psychiatry.
- [Background] Liddle, H. A. (2002). Multidimensional family therapy for adolescent cannabis users. Cannabis Youth Treatment (CYT) Series, Volume 5. Rockville: Center for Substance Abuse Treatment, Substance Abuse and Mental Health Services Administration.
- [Background] Nock, M. K., & Photos, V. (2006). Parent motivation to participate in treatment: Assessment and prediction of subsequent participation. Journal of Child and Family Studies, 15, 333-346. https://doi.org/10.1007/s10826-006-9022-4
- [Background] Tolan PH, Hanish LD, McKay MM, Dickey MH. Evaluating process in child and family interventions: aggression prevention as an example. J Fam Psychol. 2002 Jun;16(2):220-36. doi: 10.1037//0893-3200.16.2.220. PMID 12085734
- [Background] Van der Helm GH, Wissink IB, De Jongh T, Stams GJ. Measuring treatment motivation in secure juvenile facilities. Int J Offender Ther Comp Criminol. 2013 Aug;57(8):996-1008. doi: 10.1177/0306624X12443798. Epub 2012 May 23. PMID 22627687
- [Background] van der Helm, P., Kuiper, C. H. Z. , & Stams, G. J. J. M. (2018). Group climate and treatment motivation in secure residential and forensic youth care from the perspective of self determination theory. Children and Youth Services Review, 93, 339-344. https://doi.org/10.1016/j.childyouth.2018.07.028